CLINICAL TRIAL: NCT06795997
Title: ETM Taxes: The Impact of Innovative Tax Proposals on Purchase Patterns Across SES
Brief Title: Tobacco/Nicotine Purchase Patterns Across SES
Acronym: AIM2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Stein, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VT IRB 24-1228; 5R01CA266966 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2025-01-28 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Smoking Behaviors; Smoking, Non-Tobacco Products; Smoking, Cigarette
Keywords: Experimental Tobacco Marketplace; Tobacco Regulatory Policy
MeSH Terms: conditions — Smoking; Smoking, Non-Tobacco Products; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Within-subject design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exclusive Cigarette Smokers (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to all of the tax conditions described in the intervention section.
  Interventions: Behavioral: Tax Conditions
- Exclusive Cigarette Smokers-Control Condition (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to the control condition described in the intervention section.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: Tax Conditions — Participants will make hypothetical purchases of tobacco products to use throughout the next 7 days. Participants will complete a total of 21 purchasing trials each for 7 days' worth of products. They will be exposed to 4 conditions with 5 trials each, where products will increase in price: Tobacco Parity, Nicotine-Content, Harm- Reduction, and Modified Risk Tobacco Product-related taxes.
  Arms: Exclusive Cigarette Smokers
Behavioral: Control Condition — Participants will make hypothetical purchases of tobacco products to use throughout the next 7 days. Participants will complete a total of 21 purchasing trials each for 7 days' worth of products. They will be exposed to a control trial.
  Arms: Exclusive Cigarette Smokers-Control Condition

SUMMARY:
In a within-subject design, investigators will use the Experimental Tobacco Marketplace (ETM) to systematically impose 4 novel tobacco/nicotine tax proposals (Tobacco Parity, Nicotine-Content, Harm-Reduction, and Modified Risk Tobacco Product-related taxes) covering a broad range of tax magnitudes. Participants will complete one control trial and all conditions (tax proposals) in the ETM with 5 trials each. Analyses will model the quantity of the product purchased as a function of tax tier (i.e., high, medium, no tax) and examine poly-tobacco purchasing.

DETAILED DESCRIPTION:
Although taxes have been studied in econometric and quasi-experimental studies, the ETM is the only experimental laboratory model that has examined the impact of taxes on purchasing behavior. In pilot data collected originally for the prior version of this grant's application, investigators examined the Tobacco Parity Tax and Harm-Reduction Tax among exclusive cigarette smokers (n=35) in an online hypothetical ETM. Briefly, each tax proposal had 3 tax tiers (see C.1 Implementation of Tax Proposals, for the rationale) in the ETM with a subset of products. Therein, the Tobacco Parity Tax decreased purchases from the highest tax tier (p<0.001; f=0.49) and increased purchases of the no-tax tier (nicotine gum/lozenges were the most purchased; p<0.001; f=0.36) as taxes increased.

Conversely, the Harm-Reduction Tax resulted in greater purchases from the middle tier as tax constraints increased (ENDS were the most purchased; p<0.001; f=0.29). Moreover, the Harm-Reduction Tax elicited a greater substitution of medium-tiered products compared to the Tobacco Parity Tax (p<0.001; f=0.15). In follow-up secondary analyses of this preliminary data, investigators stratified these tax proposal by SES and found the largest effect in the Harm-Reduction Tax with the low SES group exhibiting the highest substitution of medium-tax tier products compared to more affluent groups (ps<0.001; f=0.16; Fig. 3). These results must be replicated with larger samples. In this study, investigators will ensure socioeconomic representation reflective of the US population. Given the robust effect of tax magnitude, investigators will also examine purchasing across a broad range of magnitudes to fully characterize each novel tax proposal-thereby discerning how smokers will defend their consumption or substitute with other products.

Participants will complete a one session study including consent and behavioral tasks (ETM and smoking-related assessments). A Qualtrics survey will administer:

1. the electronic informed consent; Participants will read through the informed consent and consent will be implied with submission of the assessment at the end of the survey.
2. smoking-related assessments

   1. timeline follow back, to assess previous month recent smoking, e-cigarette use and consumption of nicotine products, and to determine ETM budget
   2. tobacco use history, exposure and preferences questions;
   3. the Fagerstrom Test of Nicotine Dependence for cigarettes and the Heaviness of Smoking Index for e-cigarettes to assess dependence.
3. the ETM; Participants will make hypothetical purchases of tobacco products to use throughout the next 7 days. Participants will complete a total of 21 purchasing trials each for 7 days' worth of products. They will be exposed to a control trial and 4 conditions with 5 trials each, where products will increase in price: Tobacco Parity, Nicotine-Content, Harm- Reduction, and Modified Risk Tobacco Product-related taxes.

ELIGIBILITY:
Inclusion Criteria:

* provide informed consent
* be at least 21 years of age
* smoke at least 10 cigarettes daily and use other tobacco products less than weekly

Exclusion Criteria:

• pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 663 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Tobacco Product Purchasing | During a one-session study, participants will complete a total of 21 purchasing trials each for 7 days' worth of products. They will be exposed to a control trial and 4 conditions with 5 trials each, where products will increase in price
  Participants will make hypothetical purchases of tobacco products to use throughout the next 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Stein, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No